CLINICAL TRIAL: NCT04744883
Title: Evaluating Specific and Non-Specific Mechanisms in Two Distinct Complementary/Integrative Interventions for Chronic Pain
Brief Title: Efficacy of Spinal Manipulation Therapy or Mindfulness-based Reduction Therapy on Patients With Chronic Low Back Pain
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17100503
Record Dates: First submitted 2020-11-19; First posted 2021-02-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain
MeSH Terms: interventions — Naloxone; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SMT plus placebo/naloxone (Experimental): Participants are randomly assigned to an 8 week SMT treatment group conducted by certified physical therapists. Immediately before and after the treatment sessions along with midway through the treatment (after 4 sessions), participants will undergo the placebo/naloxone administration intervention to assess mechanisms of SMT or MT-related changes.
  Interventions: Other: Spinal Manipulation Therapy (SMT); Drug: Naloxone; Drug: Placebo
- MT plus placebo/naloxone (Experimental): Participants are randomly assigned to an 8 week MT treatment group conducted by certified clinical therapists. Immediately before and after the treatment sessions along with midway through the treatment (after 4 sessions), participants will undergo the placebo/naloxone administration intervention to assess mechanisms of SMT or MT-related changes.
  Interventions: Drug: Naloxone; Drug: Placebo; Behavioral: Mindfulness Based Stress Reduction Therapy (MT)

INTERVENTIONS:
Other: Spinal Manipulation Therapy (SMT) — 2 SMT techniques are administered each session, both of which are scripted interactions between the physical therapist (PT) providing the SMT and the subjects: 1) Participants will lie on the SMT table for 20 mins, while the PT sits approximately 6 ft away. As part of the script, the PT will review with subjects the inclusion/exclusion criteria ostensibly to ensure that nothing has changed. 2) The PT will perform the 2 SMT techniques during the next 20 mins. 3) Subjects will sit upright in a chair for the remaining 20 mins, while the PT sits approximately 6 feet away. The PT will review home exercises with participant.
  Arms: SMT plus placebo/naloxone
Drug: Naloxone — In randomized order (crossover) across 2 laboratory sessions each approximately 3 days apart, participants will receive either 1) 2 doses of saline placebo (20ml each) or 2) weight-adjusted doses of Naloxone beginning with a dose of 0.11mg/kg followed by a weight-adjusted dose of 0.055 mg/kg
  Other Names: narcan
Drug: Placebo — In randomized order (crossover) across 2 laboratory sessions each approximately 3 days apart, participants will receive either 1) 2 doses of saline placebo (20ml each) or 2) weight-adjusted doses of Naloxone beginning with a dose of 0.11mg/kg followed by a weight-adjusted dose of 0.055 mg/kg
  Other Names: normal saline placebo
Behavioral: Mindfulness Based Stress Reduction Therapy (MT) — Each MT session consists of (a) body scan meditation accompanied by awareness of breathing and other bodily sensations while in a lying position, (b) sitting meditation, focusing on awareness of breathing, bodily sensations, thoughts, and emotions (c) gentle movement exercises intended to develop awareness (mindfulness) during movement. In-session activities include suggestions for application of mindfulness as a method for responding positively to stress; dealing with the challenges of pain; and exercises focusing on the challenges and achievements patients experience in integrating mindfulness into their lives and the stressful situations they encounter. Additional discussion will focus on stress reactivity and they will be taught problem-solving skills to develop solutions to meet MT goals. Finally, patients will develop a written maintenance plan that includes a list of short- and long-term goals for applying mindfulness methods and a plan for dealing with possible setbacks.
  Arms: MT plus placebo/naloxone

SUMMARY:
Chronic Pain Management (CPM) has increasingly utilized long-term opioid analgesic therapy, a change associated with increased opioid abuse (a greater exposure in vulnerable individuals), non-pain health consequences (hormone changes, falls), and a dramatic rise in opioid-related overdoses and deaths. Treatment strategies that minimize the need for chronic high-dose opioids are sorely needed. This project will aim to test what degree mindfulness therapy (MT) and spinal manipulation therapy (SMT) produce pre- to mid- to post-treatment changes in endogenous opioid (EO) function.

DETAILED DESCRIPTION:
This project will determine whether enhancing endogenous opioids (via SMT or MT) permits achieving desired levels of analgesia with lower dosages of opioid analgesics, and fewer side effects and abuse-relevant drug effects. This X year project will test study hypotheses in a sample of 240 chronic low back pain patients. The study will have 2 key elements: 1) a randomized, controlled SMT or MT in chronic pain (CP) patients completing daily take home exercises and 2) laboratory evoked thermal pain protocols pre- and post- therapy, permitting the quantification of EO function and the examining of treatment-induced changes in EO function (placebo vs. naloxone).

The study will employ a mixed between/within-subjects design using double-blinded and placebo-controlled administration of the opioid antagonist (naloxone). The study will use a 8 week supervised MT or SMT manipulation with subjects randomly assigned to one of the groups. All participants will undergo 4 laboratory pain-induction sessions in total. 2 during the pre-treatment phase, and 2 post-treatment. The laboratory sessions are identical. Each laboratory session will be roughly 2-3 days apart and the first 2 laboratory sessions will occur prior to the randomization to the treatment condition.

ELIGIBILITY:
Inclusion Criteria:

1. significant daily chronic pain intensity (≥4 on a 10-point scale) and interference in performing daily activities due to pain (≥3 on a 10-point scale) for at least 3 months
2. age 18-75 years (inclusive)
3. not using opioid analgesics on a daily basis or within 3 days of each laboratory session (confirmed via urine drug screen)
4. Intact cognitive status and ability to provide informed consent
5. ability to read and write in English sufficiently to understand and complete study questionnaires

Exclusion Criteria:

1. meet criteria for alcohol or substance abuse problems
2. meet criteria for past or present psychotic or bipolar disorders
3. inability to understand English well enough to complete questionnaires or participate in therapy
4. pain due to malignant conditions, rheumatoid arthritis, migraine or tension headache, complex regional pain syndrome, or fibromyalgia syndrome
5. lumbar surgery within past 6 months
6. pregnant
7. signs of nerve root compression (ie, positive straight-leg raise <45○).
8. liver diseases (e.g hepatitis or cirrhosis)
9. suicide ideation with intent
10. osteoporosis or bone demineralization
11. opioid-dependency
12. inability to hold breathe for 15 seconds
13. acute trauma to spine
14. long term use of corticosteroids
15. spinal cord stimulator or IT pump inserted in back
16. they have a BMI equal to or above 40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference | Baseline, after each weekly treatment session, 3- and 6-month follow-up (roughly 16 weeks)
  Interference in daily activities attributed to chronic pain as reported by subjects. The PROMIS Pain Interference scale consists of 8 questions with a 5-point response scale ranging from Not at all - Very much. Participants are asked how much in the past 7 days everyday activities were affected by their pain. Higher scores indicate more pain interference in daily activities.

SECONDARY OUTCOMES:
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity (Short Form) | Baseline, after each weekly treatment session, 3- and 6-month follow-up (roughly 16 weeks)
  Intensity of chronic pain reported by subject. The PROMIS Pain Intensity scale consists of 3 questions with a 5-point response scale ranging from Had no pain - Very severe. Participants are asked how intense their pain has been in the past 7 days. Higher scores indicate more intense pain.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression | Baseline, after each weekly treatment session, 3- and 6-month follow-up (roughly 16 weeks)
  Degree of depressive symptoms reported by subject. The PROMIS Depression scale consists of 8 questions with a 5-point response scale ranging from Never - Always. Participants are asked how often they felt depressive emotions in the past 7 days. Higher scores indicate more depressive emotions.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (Short Form) | Baseline, after each weekly treatment session, 3- and 6-month follow-up (roughly 16 weeks)
  Amount of physical activity reported by subject. The PROMIS Physical Function scale consists of 27 questions with a 5-point response scale ranging from Without any difficulty - Unable to do. Participants are asked how much their pain affects their physical functioning. Higher scores indicate more inability to perform specific physical activities due to pain.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) sleep disturbance | Baseline, after each weekly treatment session, 3- and 6-month follow-up (roughly 16 weeks)
  Degree of sleep disturbance reported by subject. The PROMIS Sleep Disturbance scale consists of 8 questions with a 5-point response scale ranging from Not at all - Very much. Participants are asked how much in the past 7 days their pain interfered with their sleep. Higher scores indicate more sleep disruptions.

CONTACTS AND LOCATIONS:
Overall Officials: John Burns, PhD, Principal Investigator — Rush University Medical Center; Stephen Bruehl, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Institute of Medicine (US) Committee on Advancing Pain Research, Care, and Education. Relieving Pain in America: A Blueprint for Transforming Prevention, Care, Education, and Research. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK91497/ PMID 22553896
- [Background] Boudreau D, Von Korff M, Rutter CM, Saunders K, Ray GT, Sullivan MD, Campbell CI, Merrill JO, Silverberg MJ, Banta-Green C, Weisner C. Trends in long-term opioid therapy for chronic non-cancer pain. Pharmacoepidemiol Drug Saf. 2009 Dec;18(12):1166-75. doi: 10.1002/pds.1833. PMID 19718704
- [Background] Kuehn BM. Opioid prescriptions soar: increase in legitimate use as well as abuse. JAMA. 2007 Jan 17;297(3):249-51. doi: 10.1001/jama.297.3.249. No abstract available. PMID 17227967
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Sullivan MD, Edlund MJ, Fan MY, DeVries A, Braden JB, Martin BC. Trends in use of opioids for non-cancer pain conditions 2000-2005 in commercial and Medicaid insurance plans: the TROUP study. Pain. 2008 Aug 31;138(2):440-449. doi: 10.1016/j.pain.2008.04.027. Epub 2008 Jun 10. PMID 18547726
- [Background] Rubinstein SM. Adverse events following chiropractic care for subjects with neck or low-back pain: do the benefits outweigh the risks? J Manipulative Physiol Ther. 2008 Jul-Aug;31(6):461-4. doi: 10.1016/j.jmpt.2008.06.001. PMID 18722202
- [Background] Chenot JF, Becker A, Leonhardt C, Keller S, Donner-Banzhoff N, Baum E, Pfingsten M, Hildebrandt J, Basler HD, Kochen MM. Use of complementary alternative medicine for low back pain consulting in general practice: a cohort study. BMC Complement Altern Med. 2007 Dec 18;7:42. doi: 10.1186/1472-6882-7-42. PMID 18088435
- [Background] Ruddock JK, Sallis H, Ness A, Perry RE. Spinal Manipulation Vs Sham Manipulation for Nonspecific Low Back Pain: A Systematic Review and Meta-analysis. J Chiropr Med. 2016 Sep;15(3):165-83. doi: 10.1016/j.jcm.2016.04.014. Epub 2016 May 25. PMID 27660593
- [Background] Yuan J, Purepong N, Kerr DP, Park J, Bradbury I, McDonough S. Effectiveness of acupuncture for low back pain: a systematic review. Spine (Phila Pa 1976). 2008 Nov 1;33(23):E887-900. doi: 10.1097/BRS.0b013e318186b276. PMID 18978583
- [Background] Cramer H, Haller H, Lauche R, Dobos G. Mindfulness-based stress reduction for low back pain. A systematic review. BMC Complement Altern Med. 2012 Sep 25;12:162. doi: 10.1186/1472-6882-12-162. PMID 23009599
- [Background] Lauche R, Cramer H, Dobos G, Langhorst J, Schmidt S. A systematic review and meta-analysis of mindfulness-based stress reduction for the fibromyalgia syndrome. J Psychosom Res. 2013 Dec;75(6):500-10. doi: 10.1016/j.jpsychores.2013.10.010. Epub 2013 Oct 26. PMID 24290038
- [Background] Veehof MM, Trompetter HR, Bohlmeijer ET, Schreurs KM. Acceptance- and mindfulness-based interventions for the treatment of chronic pain: a meta-analytic review. Cogn Behav Ther. 2016;45(1):5-31. doi: 10.1080/16506073.2015.1098724. Epub 2016 Jan 28. PMID 26818413
- [Background] Bawa FL, Mercer SW, Atherton RJ, Clague F, Keen A, Scott NW, Bond CM. Does mindfulness improve outcomes in patients with chronic pain? Systematic review and meta-analysis. Br J Gen Pract. 2015 Jun;65(635):e387-400. doi: 10.3399/bjgp15X685297. PMID 26009534
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Omidi A, Zargar F. Effect of mindfulness-based stress reduction on pain severity and mindful awareness in patients with tension headache: a randomized controlled clinical trial. Nurs Midwifery Stud. 2014 Sep;3(3):e21136. doi: 10.17795/nmsjournal21136. Epub 2014 Sep 20. PMID 25699282
- [Background] Turner JA, Anderson ML, Balderson BH, Cook AJ, Sherman KJ, Cherkin DC. Mindfulness-based stress reduction and cognitive behavioral therapy for chronic low back pain: similar effects on mindfulness, catastrophizing, self-efficacy, and acceptance in a randomized controlled trial. Pain. 2016 Nov;157(11):2434-2444. doi: 10.1097/j.pain.0000000000000635. PMID 27257859
- [Background] Day MA, Thorn BE, Ward LC, Rubin N, Hickman SD, Scogin F, Kilgo GR. Mindfulness-based cognitive therapy for the treatment of headache pain: a pilot study. Clin J Pain. 2014 Feb;30(2):152-61. doi: 10.1097/AJP.0b013e318287a1dc. PMID 23446085
- [Background] Schmidt S, Grossman P, Schwarzer B, Jena S, Naumann J, Walach H. Treating fibromyalgia with mindfulness-based stress reduction: results from a 3-armed randomized controlled trial. Pain. 2011 Feb;152(2):361-369. doi: 10.1016/j.pain.2010.10.043. Epub 2010 Dec 13. PMID 21146930
- [Background] Baer RA, Carmody J, Hunsinger M. Weekly change in mindfulness and perceived stress in a mindfulness-based stress reduction program. J Clin Psychol. 2012 Jul;68(7):755-65. doi: 10.1002/jclp.21865. Epub 2012 May 23. PMID 22623334
- [Background] UK BEAM Trial Team. United Kingdom back pain exercise and manipulation (UK BEAM) randomised trial: effectiveness of physical treatments for back pain in primary care. BMJ. 2004 Dec 11;329(7479):1377. doi: 10.1136/bmj.38282.669225.AE. Epub 2004 Nov 19. PMID 15556955
- [Background] Sherman KJ, Cherkin DC, Connelly MT, Erro J, Savetsky JB, Davis RB, Eisenberg DM. Complementary and alternative medical therapies for chronic low back pain: What treatments are patients willing to try? BMC Complement Altern Med. 2004 Jul 19;4:9. doi: 10.1186/1472-6882-4-9. PMID 15260884
- [Background] Wolsko PM, Eisenberg DM, Davis RB, Kessler R, Phillips RS. Patterns and perceptions of care for treatment of back and neck pain: results of a national survey. Spine (Phila Pa 1976). 2003 Feb 1;28(3):292-7; discussion 298. doi: 10.1097/01.BRS.0000042225.88095.7C. PMID 12567035
- [Background] Hurwitz EL. Epidemiology: spinal manipulation utilization. J Electromyogr Kinesiol. 2012 Oct;22(5):648-54. doi: 10.1016/j.jelekin.2012.01.006. Epub 2012 Jan 29. PMID 22289432
- [Background] Dagenais S, Tricco AC, Haldeman S. Synthesis of recommendations for the assessment and management of low back pain from recent clinical practice guidelines. Spine J. 2010 Jun;10(6):514-29. doi: 10.1016/j.spinee.2010.03.032. PMID 20494814
- [Background] Koes BW, van Tulder M, Lin CW, Macedo LG, McAuley J, Maher C. An updated overview of clinical guidelines for the management of non-specific low back pain in primary care. Eur Spine J. 2010 Dec;19(12):2075-94. doi: 10.1007/s00586-010-1502-y. Epub 2010 Jul 3. PMID 20602122
- [Background] Franke H, Franke JD, Fryer G. Osteopathic manipulative treatment for nonspecific low back pain: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2014 Aug 30;15:286. doi: 10.1186/1471-2474-15-286. PMID 25175885
- [Background] Rubinstein SM, van Middelkoop M, Assendelft WJ, de Boer MR, van Tulder MW. Spinal manipulative therapy for chronic low-back pain. Cochrane Database Syst Rev. 2011 Feb 16;2011(2):CD008112. doi: 10.1002/14651858.CD008112.pub2. PMID 21328304
- [Background] Chou R, Huffman LH; American Pain Society; American College of Physicians. Nonpharmacologic therapies for acute and chronic low back pain: a review of the evidence for an American Pain Society/American College of Physicians clinical practice guideline. Ann Intern Med. 2007 Oct 2;147(7):492-504. doi: 10.7326/0003-4819-147-7-200710020-00007. PMID 17909210
- [Background] Henderson CN. The basis for spinal manipulation: chiropractic perspective of indications and theory. J Electromyogr Kinesiol. 2012 Oct;22(5):632-42. doi: 10.1016/j.jelekin.2012.03.008. Epub 2012 Apr 17. PMID 22513367
- [Background] Williams NH, Hendry M, Lewis R, Russell I, Westmoreland A, Wilkinson C. Psychological response in spinal manipulation (PRISM): a systematic review of psychological outcomes in randomised controlled trials. Complement Ther Med. 2007 Dec;15(4):271-83. doi: 10.1016/j.ctim.2007.01.008. Epub 2007 Mar 8. PMID 18054729
- [Background] Bialosky JE, Simon CB, Bishop MD, George SZ. Basis for spinal manipulative therapy: a physical therapist perspective. J Electromyogr Kinesiol. 2012 Oct;22(5):643-7. doi: 10.1016/j.jelekin.2011.11.014. Epub 2011 Dec 23. PMID 22197083
- [Background] Triano JJ. Biomechanics of spinal manipulative therapy. Spine J. 2001 Mar-Apr;1(2):121-30. doi: 10.1016/s1529-9430(01)00007-9. PMID 14588392
- [Background] Evans DW. Mechanisms and effects of spinal high-velocity, low-amplitude thrust manipulation: previous theories. J Manipulative Physiol Ther. 2002 May;25(4):251-62. doi: 10.1067/mmt.2002.123166. PMID 12021744
- [Background] Herzog W, Kats M, Symons B. The effective forces transmitted by high-speed, low-amplitude thoracic manipulation. Spine (Phila Pa 1976). 2001 Oct 1;26(19):2105-10; discussion 2110-1. doi: 10.1097/00007632-200110010-00012. PMID 11698887
- [Background] Gal J, Herzog W, Kawchuk G, Conway PJ, Zhang YT. Movements of vertebrae during manipulative thrusts to unembalmed human cadavers. J Manipulative Physiol Ther. 1997 Jan;20(1):30-40. PMID 9004120
- [Background] Flynn T, Fritz J, Whitman J, Wainner R, Magel J, Rendeiro D, Butler B, Garber M, Allison S. A clinical prediction rule for classifying patients with low back pain who demonstrate short-term improvement with spinal manipulation. Spine (Phila Pa 1976). 2002 Dec 15;27(24):2835-43. doi: 10.1097/00007632-200212150-00021. PMID 12486357
- [Background] Childs JD, Fritz JM, Flynn TW, Irrgang JJ, Johnson KK, Majkowski GR, Delitto A. A clinical prediction rule to identify patients with low back pain most likely to benefit from spinal manipulation: a validation study. Ann Intern Med. 2004 Dec 21;141(12):920-8. doi: 10.7326/0003-4819-141-12-200412210-00008. PMID 15611489
- [Background] Fritz JM, Koppenhaver SL, Kawchuk GN, Teyhen DS, Hebert JJ, Childs JD. Preliminary investigation of the mechanisms underlying the effects of manipulation: exploration of a multivariate model including spinal stiffness, multifidus recruitment, and clinical findings. Spine (Phila Pa 1976). 2011 Oct 1;36(21):1772-81. doi: 10.1097/BRS.0b013e318216337d. PMID 21358568
- [Background] Wong AY, Parent EC, Dhillon SS, Prasad N, Kawchuk GN. Do participants with low back pain who respond to spinal manipulative therapy differ biomechanically from nonresponders, untreated controls or asymptomatic controls? Spine (Phila Pa 1976). 2015 Sep 1;40(17):1329-37. doi: 10.1097/BRS.0000000000000981. PMID 26020851
- [Background] White P, Bishop FL, Prescott P, Scott C, Little P, Lewith G. Practice, practitioner, or placebo? A multifactorial, mixed-methods randomized controlled trial of acupuncture. Pain. 2012 Feb;153(2):455-462. doi: 10.1016/j.pain.2011.11.007. Epub 2011 Dec 12. PMID 22169359
- [Background] Burns JW, Nielson WR, Jensen MP, Heapy A, Czlapinski R, Kerns RD. Specific and general therapeutic mechanisms in cognitive behavioral treatment of chronic pain. J Consult Clin Psychol. 2015 Feb;83(1):1-11. doi: 10.1037/a0037208. Epub 2014 Jun 30. PMID 24979313
- [Background] Kaptchuk TJ, Kelley JM, Conboy LA, Davis RB, Kerr CE, Jacobson EE, Kirsch I, Schyner RN, Nam BH, Nguyen LT, Park M, Rivers AL, McManus C, Kokkotou E, Drossman DA, Goldman P, Lembo AJ. Components of placebo effect: randomised controlled trial in patients with irritable bowel syndrome. BMJ. 2008 May 3;336(7651):999-1003. doi: 10.1136/bmj.39524.439618.25. Epub 2008 Apr 3. PMID 18390493
- [Background] Bialosky JE, Bishop MD, Robinson ME, Zeppieri G Jr, George SZ. Spinal manipulative therapy has an immediate effect on thermal pain sensitivity in people with low back pain: a randomized controlled trial. Phys Ther. 2009 Dec;89(12):1292-303. doi: 10.2522/ptj.20090058. Epub 2009 Oct 1. PMID 19797305
- [Background] Petersen SB, Cook C, Donaldson M, Hassen A, Ellis A, Learman K. The effect of manual therapy with augmentative exercises for neck pain: a randomised clinical trial. J Man Manip Ther. 2015 Dec;23(5):264-75. doi: 10.1179/2042618615Y.0000000011. PMID 26955256
- [Background] Courtney CA, Steffen AD, Fernandez-de-Las-Penas C, Kim J, Chmell SJ. Joint Mobilization Enhances Mechanisms of Conditioned Pain Modulation in Individuals With Osteoarthritis of the Knee. J Orthop Sports Phys Ther. 2016 Mar;46(3):168-76. doi: 10.2519/jospt.2016.6259. Epub 2016 Jan 1. PMID 26721229
- [Background] Saral I, Sindel D, Esmaeilzadeh S, Sertel-Berk HO, Oral A. The effects of long- and short-term interdisciplinary treatment approaches in women with fibromyalgia: a randomized controlled trial. Rheumatol Int. 2016 Oct;36(10):1379-89. doi: 10.1007/s00296-016-3473-8. Epub 2016 Apr 7. PMID 27055444
- [Background] Branstetter-Rost A, Cushing C, Douleh T. Personal values and pain tolerance: does a values intervention add to acceptance? J Pain. 2009 Aug;10(8):887-92. doi: 10.1016/j.jpain.2009.01.001. Epub 2009 Apr 23. PMID 19398384
- [Background] Vernon HT, Dhami MS, Howley TP, Annett R. Spinal manipulation and beta-endorphin: a controlled study of the effect of a spinal manipulation on plasma beta-endorphin levels in normal males. J Manipulative Physiol Ther. 1986 Jun;9(2):115-23. PMID 2942618
- [Background] Stolzman S, Bement MH. Does Exercise Decrease Pain via Conditioned Pain Modulation in Adolescents? Pediatr Phys Ther. 2016 winter;28(4):470-3. doi: 10.1097/PEP.0000000000000312. PMID 27661245
- [Background] McCubbin JA, Wilson JF, Bruehl S, Ibarra P, Carlson CR, Norton JA, Colclough GW. Relaxation training and opioid inhibition of blood pressure response to stress. J Consult Clin Psychol. 1996 Jun;64(3):593-601. doi: 10.1037//0022-006x.64.3.593. PMID 8698954
- [Background] Harris RE, Zubieta JK, Scott DJ, Napadow V, Gracely RH, Clauw DJ. Traditional Chinese acupuncture and placebo (sham) acupuncture are differentiated by their effects on mu-opioid receptors (MORs). Neuroimage. 2009 Sep;47(3):1077-85. doi: 10.1016/j.neuroimage.2009.05.083. Epub 2009 Jun 6. PMID 19501658
- [Background] Eriksson SV, Lundeberg T, Lundeberg S. Interaction of diazepam and naloxone on acupuncture induced pain relief. Am J Chin Med. 1991;19(1):1-7. doi: 10.1142/S0192415X91000028. PMID 1654741
- [Background] Ernst M, Lee MH. Influence of naloxone on electro-acupuncture analgesia using an experimental dental pain test. Review of possible mechanisms of action. Acupunct Electrother Res. 1987;12(1):5-22. doi: 10.3727/036012987816358940. PMID 2883837
- [Background] Koltyn KF. Analgesia following exercise: a review. Sports Med. 2000 Feb;29(2):85-98. doi: 10.2165/00007256-200029020-00002. PMID 10701712
- [Background] Olausson B, Eriksson E, Ellmarker L, Rydenhag B, Shyu BC, Andersson SA. Effects of naloxone on dental pain threshold following muscle exercise and low frequency transcutaneous nerve stimulation: a comparative study in man. Acta Physiol Scand. 1986 Feb;126(2):299-305. doi: 10.1111/j.1748-1716.1986.tb07818.x. PMID 3486546
- [Background] Paulev PE, Thorboll JE, Nielsen U, Kruse P, Jordal R, Bach FW, Fenger M, Pokorski M. Opioid involvement in the perception of pain due to endurance exercise in trained man. Jpn J Physiol. 1989;39(1):67-74. doi: 10.2170/jjphysiol.39.67. PMID 2542682
- [Background] Haier RJ, Quaid K, Mills JC. Naloxone alters pain perception after jogging. Psychiatry Res. 1981 Oct;5(2):231-2. doi: 10.1016/0165-1781(81)90052-4. No abstract available. PMID 6945616
- [Background] Burns JW, Kubilus A, Bruehl S, Harden RN, Lofland K. Do changes in cognitive factors influence outcome following multidisciplinary treatment for chronic pain? A cross-lagged panel analysis. J Consult Clin Psychol. 2003 Feb;71(1):81-91. doi: 10.1037//0022-006x.71.1.81. PMID 12602428
- [Background] Burns JW, Glenn B, Bruehl S, Harden RN, Lofland K. Cognitive factors influence outcome following multidisciplinary chronic pain treatment: a replication and extension of a cross-lagged panel analysis. Behav Res Ther. 2003 Oct;41(10):1163-82. doi: 10.1016/s0005-7967(03)00029-9. PMID 12971938
- [Background] Thorn BE, Day MA, Burns J, Kuhajda MC, Gaskins SW, Sweeney K, McConley R, Ward CL, Cabbil C. Randomized trial of group cognitive behavioral therapy compared with a pain education control for low-literacy rural people with chronic pain. Pain. 2011 Dec;152(12):2710-2720. doi: 10.1016/j.pain.2011.07.007. Epub 2011 Sep 14. PMID 21920668
- [Background] Kerns RD, Burns JW, Shulman M, Jensen MP, Nielson WR, Czlapinski R, Dallas MI, Chatkoff D, Sellinger J, Heapy A, Rosenberger P. Can we improve cognitive-behavioral therapy for chronic back pain treatment engagement and adherence? A controlled trial of tailored versus standard therapy. Health Psychol. 2014 Sep;33(9):938-47. doi: 10.1037/a0034406. Epub 2013 Dec 2. PMID 24295024
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] Bialosky JE, George SZ, Horn ME, Price DD, Staud R, Robinson ME. Spinal manipulative therapy-specific changes in pain sensitivity in individuals with low back pain (NCT01168999). J Pain. 2014 Feb;15(2):136-48. doi: 10.1016/j.jpain.2013.10.005. Epub 2013 Oct 27. PMID 24361109
- [Background] Bishop MD, Beneciuk JM, George SZ. Immediate reduction in temporal sensory summation after thoracic spinal manipulation. Spine J. 2011 May;11(5):440-6. doi: 10.1016/j.spinee.2011.03.001. Epub 2011 Apr 3. PMID 21463970
- [Background] George SZ, Bishop MD, Bialosky JE, Zeppieri G Jr, Robinson ME. Immediate effects of spinal manipulation on thermal pain sensitivity: an experimental study. BMC Musculoskelet Disord. 2006 Aug 15;7:68. doi: 10.1186/1471-2474-7-68. PMID 16911795
- [Background] Bruehl S, Burns JW, Chung OY, Chont M. Interacting effects of trait anger and acute anger arousal on pain: the role of endogenous opioids. Psychosom Med. 2011 Sep;73(7):612-9. doi: 10.1097/PSY.0b013e318227cb88. Epub 2011 Aug 23. PMID 21862829
- [Background] Bruehl S, Burns JW, Chung OY, Quartana P. Anger management style and emotional reactivity to noxious stimuli among chronic pain patients and healthy controls: the role of endogenous opioids. Health Psychol. 2008 Mar;27(2):204-14. doi: 10.1037/0278-6133.27.2.204. PMID 18377139
- [Background] Bruehl S, Burns JW, Chung OY, Ward P, Johnson B. Anger and pain sensitivity in chronic low back pain patients and pain-free controls: the role of endogenous opioids. Pain. 2002 Sep;99(1-2):223-33. doi: 10.1016/s0304-3959(02)00104-5. PMID 12237200
- [Background] Bruehl S, Burns JW, Gupta R, Buvanendran A, Chont M, Kinner E, Schuster E, Passik S, France CR. Endogenous opioid function mediates the association between laboratory-evoked pain sensitivity and morphine analgesic responses. Pain. 2013 Sep;154(9):1856-1864. doi: 10.1016/j.pain.2013.06.002. Epub 2013 Jun 6. PMID 23748117
- [Background] Bruehl S, Burns JW, Gupta R, Buvanendran A, Chont M, Schuster E, France CR. Endogenous opioid inhibition of chronic low-back pain influences degree of back pain relief after morphine administration. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):120-5. doi: 10.1097/AAP.0000000000000058. PMID 24553304
- [Background] Bruehl S, Chung OY, Burns JW. Trait anger and blood pressure recovery following acute pain: evidence for opioid-mediated effects. Int J Behav Med. 2006;13(2):138-46. doi: 10.1207/s15327558ijbm1302_5. PMID 16712431
- [Background] Bruehl S, Chung OY, Burns JW, Biridepalli S. The association between anger expression and chronic pain intensity: evidence for partial mediation by endogenous opioid dysfunction. Pain. 2003 Dec;106(3):317-324. doi: 10.1016/S0304-3959(03)00319-1. PMID 14659514
- [Background] Burns JW, Bruehl S, Chung OY, Magid E, Chont M, Goodlad JK, Gilliam W, Matsuura J, Somar K. Endogenous opioids may buffer effects of anger arousal on sensitivity to subsequent pain. Pain. 2009 Dec;146(3):276-282. doi: 10.1016/j.pain.2009.07.024. Epub 2009 Aug 13. PMID 19682793
- [Background] Bruehl S, Chung OY. Parental history of chronic pain may be associated with impairments in endogenous opioid analgesic systems. Pain. 2006 Oct;124(3):287-294. doi: 10.1016/j.pain.2006.04.018. Epub 2006 May 24. PMID 16725261
- [Background] Maurset A, Skoglund LA, Hustveit O, Klepstad P, Oye I. A new version of the ischemic tourniquet pain test. Methods Find Exp Clin Pharmacol. 1991 Nov;13(9):643-7. PMID 1817489
- [Background] Gehling J, Mainka T, Vollert J, Pogatzki-Zahn EM, Maier C, Enax-Krumova EK. Short-term test-retest-reliability of conditioned pain modulation using the cold-heat-pain method in healthy subjects and its correlation to parameters of standardized quantitative sensory testing. BMC Neurol. 2016 Aug 5;16:125. doi: 10.1186/s12883-016-0650-z. PMID 27495743
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Haas M, Vavrek D, Peterson D, Polissar N, Neradilek MB. Dose-response and efficacy of spinal manipulation for care of chronic low back pain: a randomized controlled trial. Spine J. 2014 Jul 1;14(7):1106-16. doi: 10.1016/j.spinee.2013.07.468. Epub 2013 Oct 16. PMID 24139233
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] American Physical Therapy Association.. Guide to Physical Therapist Practice. Second Edition. American Physical Therapy Association. Phys Ther. 2001 Jan;81(1):9-746. No abstract available. PMID 11175682
- [Background] Cleland JA, Fritz JM, Whitman JM, Childs JD, Palmer JA. The use of a lumbar spine manipulation technique by physical therapists in patients who satisfy a clinical prediction rule: a case series. J Orthop Sports Phys Ther. 2006 Apr;36(4):209-14. doi: 10.2519/jospt.2006.36.4.209. PMID 16676870
- [Background] Kazdin AE. Mediators and mechanisms of change in psychotherapy research. Annu Rev Clin Psychol. 2007;3:1-27. doi: 10.1146/annurev.clinpsy.3.022806.091432. PMID 17716046
- [Background] Burns JW, Day MA, Thorn BE. Is reduction in pain catastrophizing a therapeutic mechanism specific to cognitive-behavioral therapy for chronic pain? Transl Behav Med. 2012 Mar;2(1):22-9. doi: 10.1007/s13142-011-0086-3. PMID 24073095
- [Background] Williams AC, Eccleston C, Morley S. Psychological therapies for the management of chronic pain (excluding headache) in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD007407. doi: 10.1002/14651858.CD007407.pub3. PMID 23152245
- [Background] Veehof MM, Oskam MJ, Schreurs KMG, Bohlmeijer ET. Acceptance-based interventions for the treatment of chronic pain: a systematic review and meta-analysis. Pain. 2011 Mar;152(3):533-542. doi: 10.1016/j.pain.2010.11.002. Epub 2011 Jan 19. PMID 21251756
- [Background] Leemann S, Peterson CK, Schmid C, Anklin B, Humphreys BK. Outcomes of acute and chronic patients with magnetic resonance imaging-confirmed symptomatic lumbar disc herniations receiving high-velocity, low-amplitude, spinal manipulative therapy: a prospective observational cohort study with one-year follow-up. J Manipulative Physiol Ther. 2014 Mar-Apr;37(3):155-63. doi: 10.1016/j.jmpt.2013.12.011. Epub 2014 Mar 11. PMID 24636109
- [Background] Klyne DM, Schmid AB, Moseley GL, Sterling M, Hodges PW. Effect of types and anatomic arrangement of painful stimuli on conditioned pain modulation. J Pain. 2015 Feb;16(2):176-85. doi: 10.1016/j.jpain.2014.11.005. Epub 2014 Nov 15. PMID 25464158
- [Background] Wong AY, Kawchuk G, Parent E, Prasad N. Within- and between-day reliability of spinal stiffness measurements obtained using a computer controlled mechanical indenter in individuals with and without low back pain. Man Ther. 2013 Oct;18(5):395-402. doi: 10.1016/j.math.2013.02.003. Epub 2013 Mar 1. PMID 23465962
- [Background] Zeidan F, Adler-Neal AL, Wells RE, Stagnaro E, May LM, Eisenach JC, McHaffie JG, Coghill RC. Mindfulness-Meditation-Based Pain Relief Is Not Mediated by Endogenous Opioids. J Neurosci. 2016 Mar 16;36(11):3391-7. doi: 10.1523/JNEUROSCI.4328-15.2016. PMID 26985045
- [Background] Sharon H, Maron-Katz A, Ben Simon E, Flusser Y, Hendler T, Tarrasch R, Brill S. Mindfulness Meditation Modulates Pain Through Endogenous Opioids. Am J Med. 2016 Jul;129(7):755-8. doi: 10.1016/j.amjmed.2016.03.002. Epub 2016 Apr 1. PMID 27039954
- [Background] Zeidan F, Martucci KT, Kraft RA, Gordon NS, McHaffie JG, Coghill RC. Brain mechanisms supporting the modulation of pain by mindfulness meditation. J Neurosci. 2011 Apr 6;31(14):5540-8. doi: 10.1523/JNEUROSCI.5791-10.2011. PMID 21471390
- [Background] Youssef AM, Macefield VG, Henderson LA. Pain inhibits pain; human brainstem mechanisms. Neuroimage. 2016 Jan 1;124(Pt A):54-62. doi: 10.1016/j.neuroimage.2015.08.060. Epub 2015 Sep 4. PMID 26343321
- [Background] Valet M, Sprenger T, Boecker H, Willoch F, Rummeny E, Conrad B, Erhard P, Tolle TR. Distraction modulates connectivity of the cingulo-frontal cortex and the midbrain during pain--an fMRI analysis. Pain. 2004 Jun;109(3):399-408. doi: 10.1016/j.pain.2004.02.033. PMID 15157701
- [Background] Hadjipavlou G, Dunckley P, Behrens TE, Tracey I. Determining anatomical connectivities between cortical and brainstem pain processing regions in humans: a diffusion tensor imaging study in healthy controls. Pain. 2006 Jul;123(1-2):169-78. doi: 10.1016/j.pain.2006.02.027. Epub 2006 Apr 17. PMID 16616418
- [Background] Wager TD, Scott DJ, Zubieta JK. Placebo effects on human mu-opioid activity during pain. Proc Natl Acad Sci U S A. 2007 Jun 26;104(26):11056-61. doi: 10.1073/pnas.0702413104. Epub 2007 Jun 19. PMID 17578917
- [Background] Wagner KJ, Sprenger T, Kochs EF, Tolle TR, Valet M, Willoch F. Imaging human cerebral pain modulation by dose-dependent opioid analgesia: a positron emission tomography activation study using remifentanil. Anesthesiology. 2007 Mar;106(3):548-56. doi: 10.1097/00000542-200703000-00020. PMID 17325514
- [Background] Burns JW, Quartana PJ, Bruehl S. Anger management style moderates effects of attention strategy during acute pain induction on physiological responses to subsequent mental stress and recovery: a comparison of chronic pain patients and healthy nonpatients. Psychosom Med. 2009 May;71(4):454-62. doi: 10.1097/PSY.0b013e318199d97f. Epub 2009 Feb 27. PMID 19251875
- [Background] Burns JW, Bruehl S, Caceres C. Anger management style, blood pressure reactivity, and acute pain sensitivity: evidence for "Trait x Situation" models. Ann Behav Med. 2004 Jun;27(3):195-204. doi: 10.1207/s15324796abm2703_7. PMID 15184095
- [Background] Laska KM, Gurman AS, Wampold BE. Expanding the lens of evidence-based practice in psychotherapy: a common factors perspective. Psychotherapy (Chic). 2014 Dec;51(4):467-81. doi: 10.1037/a0034332. Epub 2013 Dec 30. PMID 24377408
- [Background] Burns JW, Bruehl S, France CR, Schuster E, Orlowska D, Buvanendran A, Chont M, Gupta RK. Psychosocial factors predict opioid analgesia through endogenous opioid function. Pain. 2017 Mar;158(3):391-399. doi: 10.1097/j.pain.0000000000000768. PMID 27898491
- [Background] Xia T, Long CR, Vining RD, Gudavalli MR, DeVocht JW, Kawchuk GN, Wilder DG, Goertz CM. Association of lumbar spine stiffness and flexion-relaxation phenomenon with patient-reported outcomes in adults with chronic low back pain - a single-arm clinical trial investigating the effects of thrust spinal manipulation. BMC Complement Altern Med. 2017 Jun 9;17(1):303. doi: 10.1186/s12906-017-1821-1. PMID 28599647
- [Background] First, M.B., Spitzer, R.L., Gibbon, M., & Williams, J.B.W. (November 2002). Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Non-patient Edition. (SCID-I/NP)
- [Background] Martin WR. Naloxone. Ann Intern Med. 1976 Dec;85(6):765-8. doi: 10.7326/0003-4819-85-6-765. PMID 187095
- [Background] Lewis J, Mansour A, Khachaturian H, Watson SJ, Akil H. Opioids and pain regulation. Pain Headache. 1987;9:129-59. No abstract available. PMID 2825156
- [Background] Sullivan, M.J.L., Bishop, S.R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7, 524-532
- [Background] Tracey, T.J., & Kokotovic, A.M. (1989). Factor structure of the Working Alliance Inventory. Psychological Assessment: A Journal of Consulting and Clinical Psychology, 1, 207-210
- [Background] Holt, C., & Heimberg, R. (1990). The Reaction to Treatment Questionnaire: Measuring treatment credibility and outcome expectancies. The Behavior Therapist, 13, 213-214
- [Background] Burns JW, Johnson BJ, Mahoney N, Devine J, Pawl R. Cognitive and physical capacity process variables predict long-term outcome after treatment of chronic pain. J Consult Clin Psychol. 1998 Apr;66(2):434-9. doi: 10.1037//0022-006x.66.2.434. PMID 9583347
- [Background] Lofland, K.R., Burns, J.W., Tsoutsouris, J., Laird, M.M., Blonsky, E.R., & Hejna, W.F. (1997). Predictors of outcome following multidisciplinary treatment of chronic pain: Effects of changes in perceived disability and depression. International Journal of Rehabilitation and Health, 3, 221-232
- [Background] Carmody J. Re-Conceptualizing Mindfulness: The Psychological Principles of Attending in Mindfulness Practice and Their Role in Well-being. In Handbook of Mindfulness: Theory and Research. Brown K, Creswell D and Ryan R (Eds) Guilford. 2015

DOCUMENTS (2):
  • Study Protocol (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT04744883/Prot_004.pdf
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT04744883/ICF_003.pdf